CLINICAL TRIAL: NCT05181488
Title: A Prospective, Phase II Study Evaluating the Efficacy of Intraoperative Radiotherapy After Neoadjuvant Chemotherapy in Patients With Resectable Pancreatic Cancer
Brief Title: Intraoperative Radiation Therapy for Resectable Pancreatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yona Cho (Other)
Responsible Party: Sponsor-Investigator, Yona Cho, Assistant Professor, Gangnam Severance Hospital
Organization: Gangnam Severance Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2020-0038
Record Dates: First submitted 2021-12-05; First posted 2022-01-06 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Resectable Pancreatic Cancer
Keywords: Pancreatic cancer; Intraoperative radiotherapy; neoadjuvant chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention: intraoperative radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IORT group (Experimental): Intraoperative radiation therapy of 10 Gy delivered during surgery followed by adjuvant gemcitabine chemotherapy
  Interventions: Radiation: intraoperative radiotherapy, IORT

INTERVENTIONS:
Radiation: intraoperative radiotherapy, IORT — A dose of 10 Gy is prescribed to be irradiated at a depth of 5 mm from the surface of the applicator, and the radiation oncologist determines the exact irradiation time. The irradiation time may take 20 to 60 minutes depending on the size of the applicator, and the exact irradiation time is calculated after checking the quality assurance of the radiation generator before treatment every day.

SUMMARY:
This phase II study is designed to investigate the efficacy of intraoperative radiotherapy after neoadjuvant chemotherapy in patients with resectable pancreatic cancer. The purpose of the study is to show the local recurrence rate after neoadjuvant chemotherapy and IORT is superior to that of surgical resection alone from the historical control. A total of 80 patients will be enrolled, and these patients will receive IORT of 10 Gy at 5 millimeter depth of the tumor bed, following neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed with adenocarcinoma of the pancreas or clinically diagnosed with imaging examinations or tumor markers
* 20 years or older
* Performance status 0-2 based on Eastern Cooperative Oncology Group (ECOG)
* Patients with surgically resectable or borderline resectable and advanced pancreatic cancer that can be resected after neoadjuvant chemotherapy
* Patients who voluntarily decided to participate in this clinical study and signed a written informed consent

Exclusion Criteria:

* History of previous abdominal irradiation.
* When the treatment area is not included in the appropriate radiation field according to the judgment of the radiation oncologist or Durgeon
* Distant metastasis
* Other systemic conditions that, under the judgment of the attending physician, would be difficult to undergo surgery or radiiotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
3-year local recurrence rate | 3 year after intraoperative radiotherapy
  A local recurrence is defined as reappearance of cancer in the ipsilateral preserved breast or chest wall.
  The 3-year local recurrence rate is calculated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
post-operative complication | 3 year after intraoperative radiotherapy
  Evaluation of safety, including adverse events, was performed by the Principal Investigator and delegated participating investigators in the Department of Surgery and Radiation Oncology outpatient clinic.
  Toxicity is evaluated within 3 months (acute) and thereafter (chronic) after surgery, and it is performed through a questionnaire and physical examination at every visit up to 1 year after surgery and recorded.
disease free survival | 1 year and 2 year after intraoperative radiotherapy.
  Disease-free survival is defined as the time from intraoperative radiotherapy to recurrence of tumor, death or last patient contact.
Overall survival | 1 year and 2 year after intraoperative radiotherapy.
  Overall survival was defined as the time from intraoperative radiotherapy to death or last patient contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea